CLINICAL TRIAL: NCT06750380
Title: Comparative Effects of Mackenzie and Tailored Mat Exercises on Pain, Function and Disability in Post-Menopausal Women With Chronic Nonspecific Low Back Pain
Brief Title: Effects of Mackenzie and Tailored Mat Exercises in Post-Menopausal Women With Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0527
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Back Pain, Low
Keywords: exercises; disability; postmenopausal; women; chronic; low back pain
MeSH Terms: conditions — Low Back Pain; Motor Activity; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tailored mat exercise program (Experimental): The Group A will receive TENS plus moist hot pack and follow the Tailored mat exercise program for 10 weeks, two times per week, in 45-min sessions under supervision of trained physical therapist. The choice of exercises will be made based on the suggested exercises of Wood for the treatment of back pain, while the easiest versions of each exercise would be selected in order for the program to be adapted to older adults. Patient's outcomes will be measured at baseline and after 10 weeks.
  Interventions: Other: Tailored mat exercise program
- McKenzie exercises (Active Comparator): The Group B will receive McKenzie exercises plus moist hot pack and TENS in the region of lumbar spine for 10 minutes and Mckenzie exercises of seven to ten repetitions for 45 min/session two times per week for ten weeks. Patient's outcomes will be measured at baseline and after 10 weeks
  Interventions: Other: McKenzie exercises

INTERVENTIONS:
Other: Tailored mat exercise program — The Group A will receive TENS plus moist hot pack and follow the Tailored mat exercise program for 10 weeks, two times per week, in 45-min sessions under supervision of trained physical therapist. The choice of exercises will be made based on the suggested exercises of Wood for the treatment of back pain, while the easiest versions of each exercise would be selected in order for the program to be adapted to older adults. Patient's outcomes will be measured at baseline and after 10 weeks.
  Arms: Tailored mat exercise program
Other: McKenzie exercises — The Group B will receive McKenzie exercises plus moist hot pack and TENS in the region of lumbar spine for 10 minutes and Mckenzie exercises of seven to ten repetitions for 45 min/session two times per week for ten weeks. Patient's outcomes will be measured at baseline and after 10 weeks.
  Arms: McKenzie exercises

SUMMARY:
Group A will receive tailored mat exercises. Group B will receive Mckenzie exercises. A baseline treatment including moist hot pack and TENS will be given to both of these groups. All these sessions will be of 45 minutes for 2 session per week for 10 weeks.

DETAILED DESCRIPTION:
Exercise has been shown to reduce pain and improve function levels in postmenopausal women with chronic NSLBP. McKenzie method is a well-known method used in the treatment of LBP. Another method of therapeutic exercise that has shown some positive results is the Pilates method. Existing research shows that Pilates in adult women with chronic NSLBP reduces pain and disability and improves the quality of life. However, the effect of Pilates and Mckenzie exercises in postmenopausal women with chronic NSLBP remains under investigation. This study aims to examine comparative effects of Mackenzie and tailored mat exercises on pain, function and disability in post-menopausal women with chronic nonspecific low back pain and will help in providing improvements in pain and disability and hence better quality of life.

This will be a randomized Clinical trial conducted on 62 participants. Data will be collected from Combined Military Hospital Lahore, by using non-probability convenience sampling technique. Postmenopausal Women between the age of 55 to 85 with Chronic NSLBP for more than 12 weeks, a physician referral for exercise, a pain VAS score>30 mm and≤70 mm, and (TUG) test score>15 will be included in this study. Participants who are frailer, have radicular referred leg pain, radiculopathy, low back pain due to a serious pathology participation in another lower back specific exercise program in the last 6 months, participation in a previous Pilates exercise program, neurodegenerative disease, recent stroke, and cognitive impairment (Mini Mental State Exam score < 24) will be excluded from this study. A sample of 62 will be divided into two groups with 31participants in each group. Group A will receive tailored mat exercises. Group B will receive Mckenzie exercises. A baseline treatment including moist hot pack and TENS will be given to both of these groups. All these sessions will be of 45 minutes for 2 session per week for 10 weeks. Primary outcomes included will be visual analog scale (VAS) for pain, Roland-Morris Disability Questionnaire (RMDQ), timed up-and-go (TUG), at baseline, 10 weeks, and 6 months post-interventions. Data will be analyzed by using SPSS version 26.0.

ELIGIBILITY:
Inclusion Criteria:

* chronic nonspecific low back pain (more than 12 weeks)
* Moderate pain VAS>30mm and< 70mm
* TUG score of < 15s
* Female who had entered menopause (menstrual periods have stopped for 12 months)
* Stable vital signs (patient is stable and vital signs are within normal limits)
* Multigravida

Exclusion Criteria:

* Frailer individuals
* Radiculopathy (signs of sensory loss, muscle weakness, reduced tendon reflexes)
* Women suffering from pathological conditions for example cardiac disease, cancer, vertebral fracture, osteomyelitis, Rheumatoid arthritis, cauda equina syndrome) participation in another lower back specific exercise program in the last 6 months
* Participation in a previous Pilates exercise program
* Neurodegenerative disease (e.g., Parkinson's disease)
* Recent stroke and cognitive impairment (Mini Mental State Exam score < 24)
* History of recent fracture

Ages: 55 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — post-menopausal women
Enrollment: 62 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Visual analogue Scale | 10th week
  Pain experienced in the last 24 h will be assessed with the pain VAS. The scale is an unnumbered 100 mm line, one end of which has the phrase "no pain" and the other "maximum pain". A mark is placed by the patient at a point representing their pain level. That mark is then measured by the tester with a millimeter ruler. Each measurement of the pain VAS corresponded to pain experienced in the last week, with lower values indicating less pain. The pain VAS is the most commonly used instrument for measuring low back pain intensity and its use is indicated in older adults It has high reliability with an intraclass correlation coefficient (ICC) of 0.99.
Roland-Morris disability questionnaire (RMDQ) | 10th week
  Roland-Morris disability questionnaire (RMDQ) The Greek version of the RMDQ was used to assess disability associated with low back pain in the last 24 h. This questionnaire has shown high test-retest reliability in older adults, with an intraclass correlation coefficient (ICC) of 0.85. The RMDQ consists of 24 items related to the daily activities patients often report having difficulty performing due to low back pain. Every positive answer earns one point; the final score is the total sum. The higher the score, the greater is the limitation
Timed up-and-go (TUG) test | 10th week
  The TUG is a performance-based measure of functional mobility initially developed to identify mobility and balance impairments in older adults. The TUG has demonstrated high interrater and intrarater reliability when used to examine older adults (ICC=0. 99). The patient is scored based on the time required to perform the following sequence of actions: stand up from a chair, walk at their own pace a distance of 3 m to a marked spot on the floor, turn around, return to the chair and sit back down

CONTACTS AND LOCATIONS:
Overall Officials: hina gul, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- CMH (Combined Military Hospital), Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fonseca LS, Silva JP, Souza MB, Mascarenhas RO, Silva HJ, Campos MGM, Pereira LSM, Oliveira MX, Oliveira VC. Efficacy of pharmacological and non-pharmacological therapy on pain intensity and disability of older people with chronic nonspecific low back pain: a protocol for a network meta-analysis. Syst Rev. 2023 Nov 7;12(1):205. doi: 10.1186/s13643-023-02369-0. PMID 37936147
- [Background] Bais A, Mishra SA, Darda PP, Phansopkar P. Impact of 6 weeks pilates training on menopause specific symptoms and quality of life in menopausal women: a case report. Journal of Pharmaceutical Research International. 2021 Jul 19;33(37B):83-9.
- [Background] Chiarotto A, Koes BW. Nonspecific Low Back Pain. N Engl J Med. 2022 May 5;386(18):1732-1740. doi: 10.1056/NEJMcp2032396. No abstract available. PMID 35507483
- [Background] Ravindran AK, Javed J, Parthiban R, Sherrif B. Effectiveness of aerobic exercise versus pilates in postmenopausal women with non-specific chronic low back pain. Indian Journal of Physiotherapy & Occupational Therapy Print-(ISSN 0973-5666) and Electronic-(ISSN 0973-5674). 2022 Apr 13;16(2):1-8.
- [Background] Belli G, Esposito C, Campanella M, Vista E, Pegreffi F, Maietta Latessa P. Comparison of Core Stability versus McKenzie Exercises in people with low back pain: effects induced by 4 weeks of training on pain, flexibility and spine mobility. SPORT SCIENCES FOR HEALTH (ONLINE). 2022:45-.
- [Background] Stevans JM, Delitto A, Khoja SS, Patterson CG, Smith CN, Schneider MJ, Freburger JK, Greco CM, Freel JA, Sowa GA, Wasan AD, Brennan GP, Hunter SJ, Minick KI, Wegener ST, Ephraim PL, Friedman M, Beneciuk JM, George SZ, Saper RB. Risk Factors Associated With Transition From Acute to Chronic Low Back Pain in US Patients Seeking Primary Care. JAMA Netw Open. 2021 Feb 1;4(2):e2037371. doi: 10.1001/jamanetworkopen.2020.37371. PMID 33591367